CLINICAL TRIAL: NCT03931525
Title: Effect of Fractional Radiofrecuency Associated Cosmetology Derug Delivery in Treatment of Strech Marks
Brief Title: Effect of Radiofrecuency on Stretch Marks
Acronym: FRF
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Dissolution of the research team
Sponsor: Quiropraxia y Equilibrio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8042019
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Stretch Marks
Keywords: Stretch Marks; Skin Disease; Diathermy; Drug Delivery Systems
MeSH Terms: conditions — Striae Distensae; Skin Diseases; Fever | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Radiofrequency therapy with drug delivery 30 days interval (Experimental): Group that will be treated with Fractional Radiofrequency plus a regerative drug at the Gluteus or Abdomen level during 4 sessions with an interval of 30 days.
  Interventions: Device: Fractitional Radiofrecuency with Drug Delivery
- Radiofrequency Therapy without drug delivery 30 days interval (Active Comparator): Group that will be treated with Fractional Radiofrequency at the Gluteus or Abdomen level during 4 sessions with an interval of 30 days.
  Interventions: Device: Fractitional Radiofrecuency
- Radiofrequency therapy with drug delivery 15 days (Experimental): Group that will be treated with Fractional Radiofrequency plus a regerative drug at the Gluteus or Abdomen level during 4 sessions with an interval of 15 days.
  Interventions: Device: Fractitional Radiofrecuency with Drug Delivery
- Radiofrequency therapy without drug delivery 15 days (Active Comparator): Group that will be treated with Fractional Radiofrequency at the Gluteus or Abdomen level during 4 sessions with an interval of 15 days.
  Interventions: Device: Fractitional Radiofrecuency

INTERVENTIONS:
Device: Fractitional Radiofrecuency with Drug Delivery — Electromagnetic energy within the spectrum of radio frequencies applied to the skin whose purpose is to generate thermal effects and which will be complemented with a skin drug
  Arms: Radiofrequency therapy with drug delivery 15 days; Radiofrequency therapy with drug delivery 30 days interval
Device: Fractitional Radiofrecuency — Electromagnetic energy within the spectrum of radio frequencies applied to the skin whose purpose is to generate thermal effects
  Arms: Radiofrequency Therapy without drug delivery 30 days interval; Radiofrequency therapy without drug delivery 15 days

SUMMARY:
This study aims to explore the effects of fractional Radiofrecuency (RF), as well as demonstrate the performance of the new semi-ablative radiofrequency model in the treatment of stretch marks. This research is a randomized, controlled clinical trial where 32 female patients complaining of glutes and / or abdomen striations. The participants were divided into two equal groups, G1 and G2. G1 will be treated at 30-day intervals, and subdivided into 2 subgroups: G1A, 8 patients with striations in the abdomen; and G1B, 8 patients with gluteal striations. The G1A and G1B groups will be divided into 2 subgroups of 4 people each, where one group will be treated with Fractional RF associated to drug delivery, and the other group, with only Fractional RF, without the application of drug delivery. The same rule of subdivisions will occur in G2, G2A and G2B, however, the interval between applications will be every 15 days. The treatment area will be divided into a rectangle 10cm high by 10cm wide. For evaluation, the contralateral side will be used as a control, using Photogrammetry and histological analysis as a resource, which will be collected through the punch skin fragment of the infraumbilical and gluteal region, performed by a specialized physician.

DETAILED DESCRIPTION:
1. INTRODUCTION

   Stretch marks are characterized by common dermatological conditions, being aesthetically unpleasant, disturbing especially women of different age groups. Analyzing the histological aspect, they present as atrophic lesions that disperse collagen and elastic tissue, in addition to reducing the presence of skin cells such as keratinocytes, melanocytes and fibroblasts.

   It is noted that the striations may be distributed locally or numerously, disposed parallel to one another and perpendicular to the skin cleavage lines. At the beginning, the striae appear erythematous-violet, thin and may generate pruritus, characterizing its inflammatory phase.

   When the inflammatory phase passes, the striations develop into an atrophic condition, they acquire a whitish appearance, almost pearly, becoming wider, due to the rupture of elastic and collagen fibers.

   Dermatofunctional physiotherapy already has several resources to treat these effects, such as therapeutic ultrasound, cryolipolysis, radiofrequency, low intensity laser and high intensity focused ultrasound. RF heating is commonly used to cause shrinkage of dermal collagen and induce stimulation of fibroblast cells that produce a new collagen.

   Radiofrequency is a non-invasive treatment, which leads to better circulatory and nutrient supply, tissue hydration, increased oxygenation, acceleration of elimination of catabolites, lipolysis, contraction of the connective tissue promoting reorientation of collagen fibers and increase in as well as soft tissue regeneration, and is indicated for patients with mild to moderate skin flaccidity, to improve the facial and body contour, to attenuate furrows and ridges, to moderate retraction of the fibers, and to increase the thickness and density of the epithelial tissue. sub-mental area and neck and treatment of gynoid lipodystrophy, like all equipment of deep thermo therapy, causes a great cellular excitation, leading to an accentuated caloric expenditure, while we will be promoting an expressive improvement of localized fat or cellulite in the circulatory part promoting a important vasodilatation, but when there is fibrosis very early, rapid preheating with radiofrequency is recommended initially.

   Fractional RF is another possibility for the treatment of cutaneous aging. It is a procedure that emits waves that reach the deeper layers of the skin, generating energy and strong heat, but keeping the surface cooled and protected. the procedure reaches the depth of 100 microns, that is, it reaches the papillary dermis, where it causes ablation and coagulation of surrounding proteins by residual thermal damage. This both leads to contraction of existing collagen fibers and stimulates the formation of new fibers, making them more efficient in supporting the skin.

   After discovering the advantages of fractionation applied to some forms of light for skin rejuvenation, several other researches have been done, and today we have different types of laser, radiofrequency and infrared devices that use this property as a way to keep treatments safer and effective. The development of RF fractionation was then initiated. In the fractured form this feature can be used ablatively and sub ablatively, where tissues suffer less trauma.

   There is still a lot to be studied about this new therapeutic resource, and the literature on the subject is very scarce. For this reason, this research aims to elucidate and increase the knowledge about Fractional RF. Through histological analysis and other data, we seek to ensure and clarify the effects of Fractional Radiofrequency at the dermal and epidermal level.
2. GENERAL OBJECTIVE:

   -Investigate the effects of Fractional Radiofrequency in the treatment of striae of the abdominal and gluteal regions associated or not with the active permeation (Drug Delivery).
3. SPECIFIC OBJECTIVES:

   * Compare the effects of Fractional Radiofrequency on the dermal tissue in the abdominal and gluteal regions of women, associated or not with the drug permeation (Drug Delivery), through the histological analysis.
   * Demonstrate the performance of Fractional Radiofrequency equipment in the treatment of stretch marks in the abdominal and gluteal regions of women in different treatment periods (15 and 30 days), when or not associated with drug delivery.
   * Identify the performance of Fractional RF equipment in the treatment of stretch marks in abdominal and gluteal regions in different treatment periods (every 15 and 30 days).
4. HYPOTHESES:

   * The application of Fractional Radiofrequency does not interfere in the treatment of stretch marks.
   * The application of Fractional Radiofrequency interferes in the treatment of stretch marks.
   * The permeation of assets associated with fractional RF interferes with the treatment of stretch marks.
   * Asset permeation associated with Fractional RF does not interfere with the treatment of stretch marks.
5. METHODOLOGY

   5.1 CHARACTERIZATION OF STUDY AND SAMPLE:

   The research is characterized as a randomized clinical trial in which 32 female volunteers will be selected, whose main complaint is the appearance of stretch marks in the abdominal area and gluteal areas.

   5.2 LOCATION OF THE RESEARCH:

   The participats will be assisted in an outpatient dermatological and physiotherapy treatment appropriately structured for the proposed study, containing electrical network compatible with the fractional RF equipment used, an appropriate environmental cooling system for the proper functioning of the machine, and good hygiene and lighting conditions, according to the provisions of the local Sanitary Surveillance, will be in the clinic of physiotherapy, located at Av. Antônio Basílio - Lagoa Seca / Natal-RN owned by Dr. Eneida Carreiro.

   MATERIALS:

   Fractional RF Equipment, Artis model, manufactured by Tone Derm will be used. A tape measure of the brand Fiber, a scale of the mark Glicomed, a device of Plicometria and a device of ultrasonografia of high frequency (12MHz), a punch of procedure, camera of the mark Canon. For the application of the assets will be used the Concept TI Strill Monodose Fluid manufactured by Mezzo Dermocosmetics, registered in Anvisa nº 25351.379480 / 2018-17, composed by water, Edta, Hydroxyacetophenone, 1,2 - Hexanediol, Caprylyl Glycol, Disodium Edta, Glycine Soy Glycerin, Hydrogenated Lecithin, Citric Acid, Sh-Polypeptide-5, Butylene Glycol, Cetyl Hydroxyethylcellulose, Rutin, Palmitoyl Tripeptide-1, Palmitoyl Tetrapeptide-7, Phaseolus Lunatus Seed Extract, Bulbine Frutescens Leaf Juice, Bht.

   5.3 PROCEDURE METHOD:

   During treatment the participants will be treated with fractional radiofrequency, G1 will be applied at 30-day intervals and subdivided into 2 GA groups. Abdomen with 8 patients and GB gluteal with 8 patients, the GA and GB groups were divided into 2 subgroups of 4 people each, 1 group with application of drugdelivery and 1 group without the application of drugdelivery. G2 will be applied at 15-day intervals and subdivided into 2 GC groups. Abdomen with 8 patients and gluteal GD with 8 patients, the GC and GD groups were divided into 2 subgroups of 4 people each, 1 drug application group and 1 group without the application of drug delivery. The drug consists of a solution rich in cell growth factors and the investigators will be applied after the intervention with Fractal Radiofrequency.

   The following modulation parameters will be used in the Fractional Radiofrequency equipment: Deep application mode, amplitude: 100% - ON time: 50 mseg - OFF time: 5 mseg - Pulsed mode - Pulse: 1mseg. In the gluteus and abdomen will be treated using - specific radiofrequency tips fractioned with the "fork" electrode (A distance between perforations of about 1 to 2 mm must be observed). The areas where the needle will penetrate will be cleaned with 70% alcohol before the procedure, the applications in the abdomen and gluteus will occur on the right side, the left side will not receive any radiofrequency treatment, being therefore used as a control, where later participants will be invited to treat the contralateral side.

   For the histological analysis, two patients from group G1 (abdomen and gluteus) and two patients from group G2 (abdomen and gluteus), a sample of the superficial tissue through a punch 3 mm in diameter, will be removed. The procedure will be under local anesthesia and performed by a medical plastic surgeon in order to minimize the risks.
6. RISKS AND BENEFITS OF RESEARCH:

   The Radiofrequency apparatus is registered with ANVISA, the treatment is considered safe by the FDA and duly legalized its use in Brazil. Even if it is a new technique, the researchers will be assisted by a technician responsible for the machine during the entire treatment period to avoid any technical problem.

   The risks include the use of anticoagulants and liver problems (previously questioned in the initial interview with the patient during the first evaluation). If so, the participant will be excluded from the survey. Other risks are hyperemia of the skin due to the mechanism of application of the equipment that will be smoothed by the control and questioning at the beginning of the application and the patients must be with preserved sensitivity, by having the metal applicators, it can scratch, but this will be avoided with the inspection of the device before the application and with the speed of the moderate application, if it occurs the patient would receive all the necessary care and assistance to heal. The risk of burns will be reduced by controlling the temperature.

   For the patient submitted to punch the risk is scar formation and fibrosis in the area where the skin fragment will be collected, but in order to avoid these complications the removed fragment will have the smallest possible size so that it is minimally perceptible and the procedure will be performed by physician.

   In the event of any complications, we will provide the necessary assistance, including coverage of expenses, compensation for any damages resulting from research procedures, duly substantiated by specific consultations and examinations.

   The benefits of this research are related to the improvement of the striae in the treated region. As the literature cites, as well as increasing self-esteem of it.
7. DATA ANALYSIS:

   After histological study, a statistical analysis will be performed to compare the degree of organization of the collagen and elastic fibers between the different treatment groups. A descriptive and inferential statistical analysis of the data will be performed through SPSS 19.0 (StatisticalPackage for the Social Science - Version 19.0). The normality of the date will be observed by the Kolmogorov - Smirnov (KS) test. For the comparison between groups whose parametric form data will be applied the one-way anova test for intergroup comparison. The significance level of 5% (p <0.05) will be adopted.
8. EXPECTED RESULTS:

It is expected at the end of the study that the differentiated effects for conventional and Radiofrequency equipment in the dermal tissue will be demonstrated.

This study intends to evaluate the Fractional Radiofrequency effects as well as the parameters to be used, seeking to confirm what the literature cites in relation to its physiological effects. A more detailed analysis of the whole process after the application is sought, not yet clearly described by scientific studies.

Fractional Radiofrequency is expected to increase the increase of collagen fibers, preventing the process of natural skin aging and improving the appearance of stretch marks.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 and not older than 45 years
* Presence Gluteal and Abdominal Striae.
* Stretch marks aesthetic discomfort

Exclusion Criteria:

* Malignancy.
* Metal implants or abdominal or pelvic stents
* Presence of collagen diseases.
* Alteration in the synthesis of proteins.
* Alterations of the integrity of the skin such as burns, wounds, keloids, hypertrophic scars or dermatitis.
* Intake of steroidal and nonsteroidal anti-inflammatory drugs.
* Hypocaloric diet indicated by nutritionist.
* Do not agree with the intervention protocol.

Elimination Criteria

* Non-tolerance of the intervention with electrotherapy that requires the suspension of treatment.
* Non-completion of the evaluation protocol (Attendance at all scheduled sessions).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Histological changes in stretch marks | a period of 30 days or 15 days post intervention
  Analysis with electronic microscopy of the percentage increase or decrease in the type and amount of collagen, as well as circulatory changes.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Froes Meyer, PhD, Principal Investigator — Universidade Pontiguar
Locations (1):
- Universidade Potiguar, Natal, Lagoa Nova, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandrashekar BS, Sriram R, Mysore R, Bhaskar S, Shetty A. Evaluation of microneedling fractional radiofrequency device for treatment of acne scars. J Cutan Aesthet Surg. 2014 Apr;7(2):93-7. doi: 10.4103/0974-2077.138328. PMID 25136209
- [Background] Fistonic I, Sorta Bilajac Turina I, Fistonic N, Marton I. Short time efficacy and safety of focused monopolar radiofrequency device for labial laxity improvement-noninvasive labia tissue tightening. A prospective cohort study. Lasers Surg Med. 2016 Mar;48(3):254-9. doi: 10.1002/lsm.22450. Epub 2016 Jan 8. PMID 26748986
- [Background] Gonzalez-Suarez A, Gutierrez-Herrera E, Berjano E, Jimenez Lozano JN, Franco W. Thermal and elastic response of subcutaneous tissue with different fibrous septa architectures to RF heating: numerical study. Lasers Surg Med. 2015 Feb;47(2):183-95. doi: 10.1002/lsm.22301. Epub 2015 Feb 4. PMID 25651998
- [Background] Jimenez Lozano JN, Vacas-Jacques P, Anderson RR, Franco W. Effect of fibrous septa in radiofrequency heating of cutaneous and subcutaneous tissues: computational study. Lasers Surg Med. 2013 Jul;45(5):326-38. doi: 10.1002/lsm.22146. Epub 2013 Jun 3. PMID 23733512
- [Background] Key DJ. A Preliminary Study of a Transdermal Radiofrequency Device for Body Slimming. J Drugs Dermatol. 2015 Nov;14(11):1272-8. PMID 26580877
- [Background] Caruth JC. Evaluation of the Safety and Efficacy of a Novel Radiofrequency Device for Vaginal Treatment. Surg Technol Int. 2018 Jun 1;32:145-149. PMID 29791707
- [Background] Le Louarn C. [Midface region: functional anatomy, ageing process, indications and concentric malar lift]. Ann Chir Plast Esthet. 2009 Oct;54(5):411-20. doi: 10.1016/j.anplas.2009.04.003. Epub 2009 Aug 19. French. PMID 19695761
- [Background] Sadick NS, Makino Y. Selective electro-thermolysis in aesthetic medicine: a review. Lasers Surg Med. 2004;34(2):91-7. doi: 10.1002/lsm.20013. PMID 15004818
- [Background] Weiss RA. Noninvasive radio frequency for skin tightening and body contouring. Semin Cutan Med Surg. 2013 Mar;32(1):9-17. PMID 24049924
- [Background] Casabona G et al. Radiofrequência ablativa fracionada: um estudo piloto com 20 casos para rejuvenescimento da pálpebra inferior. Surg Cosmet Dermatol 2014;6(1):505.
- [Background] Crocco, E.I.; Mantovani, P. A.;Volpini, B.M.F. Em Busca Dos Tratamentos Para Striae Rubra E Striae Alba: O Desafio Do Dermatologista. Surgical & Cosmetic Dermatology, V.4, N.4, P.332-337, 2012.